CLINICAL TRIAL: NCT01327508
Title: A Prospective, Multi-center, Randomized, Comparison Study of the TRIGEN SURESHOT™ Distal Targeting vs. Standard Targeting Instrumentation
Brief Title: TRIGEN SURESHOT™ Distal Targeting System Study
Acronym: Sureshot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary endpoint voided. Dosimeters did not capture radiation dose as expected.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-TRI-01
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Femoral Shaft Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRIGEN SURESHOT Distal Targeting (Experimental): TRIGEN SURESHOT Distal Targeting Instrumentation is utilized to find screw holes.
  Interventions: Device: TRIGEN SURESHOT Distal Targeting Instrumentation.
- Standard Nailing Instrumentation. (Active Comparator): Free-hand technique utilizes x-rays to find screw holes
  Interventions: Other: Free-hand technique

INTERVENTIONS:
Device: TRIGEN SURESHOT Distal Targeting Instrumentation. — image-guided localization system
  Other Names: SURESHOT
  Arms: TRIGEN SURESHOT Distal Targeting
Other: Free-hand technique — Free-hand technique utilizes x-rays to find screw holes.
  Arms: Standard Nailing Instrumentation.

SUMMARY:
The objective of this study is to quantitate the amount of radiation both subjects and surgeons are exposed to during intramedullary nailing of the femur using the TRIGEN SURESHOT Distal Targeting System versus Standard nailing instrumentation.

DETAILED DESCRIPTION:
The TRIGEN SURESHOT™ Distal Targeting System was designed to be an intraoperative image-guided localization system to aid with drill positioning for screws during intramedullary nailing distal interlocking. It is hypothesized that this system will aid in identification of the distal holes leading to reduced exposure to radiation. The SURESHOT System provides information to the surgeon that is used to place surgical instruments utilizing electromagnetic tracking data obtained intraoperatively. It is indicated for long bone fractures treated with intramedullary nailing in which the use of stereotactic surgery may be appropriate. The hypothesis is that using the TRIGEN SURESHOT™ Distal Targeting System will allow accurate distal locking while effectively decreasing the amount of radiation exposure compared to the standard instrumentation process.

ELIGIBILITY:
Inclusion Criteria

* Unilateral femoral shaft fracture requiring intramedullary nailing in which the use of stereotactic surgery may be appropriate.
* Subject is between 18-80 years of age.
* Subject is skeletally mature
* Subject is of legal age and capable of providing legal consent.
* Subject is suitable for current Intramedullary Nailing procedure
* Subject willing to accept randomization either to the TRIGEN SURESHOT Distal Targeting System or TRIGEN standard instrumentation.

Exclusion Criteria

* Femur shaft fracture not amenable to intramedullary nailing in which the use of sterotactic surgery may be inappropriate.
* Fracture with vascular injury (Gustilo Type IIIC) requiring repair
* Open fractures where open wound is in communication with distal targeting holes and therefore would influence duration of locking procedure (i.e. potentially no need for incisions for locking screw placement).
* Fracture of the Metaphyseal distal femur with intraarticular comminution
* Known Pathological Fracture
* Subject is a prisoner
* Operative procedure for closed fracture is scheduled for greater than 2 weeks for closed fractures
* Subject has cognitive issue/mental status conditions that preclude intramedullary nailing in the judgment of the investigator.
* Contralateral femoral shaft fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Mehta, M.D., Principal Investigator — Orthopaedic Surgery, Hospital of the University of Pennsylvania; Animesh Agarwal, M.D., Principal Investigator — UT Health Science Center, Dept of Orthopaedic; Marcus Sciadini, M.D, Principal Investigator — University of Maryland Baltimore, Department of Orthopaedics; Steven Olson, M.D., Principal Investigator — Duke University Medical Center of Orthopaedic; Chad Coles, M.D., Principal Investigator — Nova Scotia Health Authority; Richard Vlasak, M.D., Principal Investigator — Dept. of Orthopaedics & Rehab University of Florida
Locations (7):
- United States (6):
  - UC Davis Medical Center, Sacramento, California
  - Department of Orthopaedics and Rehabilitation, Gainesville, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University Hospital Trauma Service, San Antonio, Texas
- Capital District Health Authority, Halifax, Nova Scotia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRIGEN SURESHOT Distal Targeting | Standard Nailing Instrumentation.
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Unilateral femoral shaft fracture requiring treatment with intramedullary nails, in which the use of sterotactic surgery may be appropriate.
Groups:
- Total: Total of all reporting groups
Arm/Group | TRIGEN SURESHOT Distal Targeting | Standard Nailing Instrumentation. | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (19.0) | 35.3 (19.5) | 36.5 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Radiation Exposure Measurement
Description: Radiation exposure measured in two ways:
  Whole body badge TLD ring badge
Time Frame: Intraoperative
Population: Primary endpoint voided. Dosimeters did not capture radiation dose as expected.
Arm/Group | TRIGEN SURESHOT Distal Targeting | Standard Nailing Instrumentation.
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Distal Locking Time
Description: Distal locking time is defined as the period between successful nail insertion without locking and the confirmation of accurate insertion of both distal screws.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TRIGEN SURESHOT Distal Targeting | Standard Nailing Instrumentation.
Number analyzed (Participants) | 30 | 30
minutes | 12.6 (6.9) | 14.7 (8.4)

ADVERSE EVENTS:
Time Frame: Operative and immediate postoperative
Arm/Group | TRIGEN SURESHOT Distal Targeting | Standard Nailing Instrumentation.
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIGEN SURESHOT Distal Targeting (N=30) | Standard Nailing Instrumentation. (N=30)
Change out screw (Surgical and medical procedures) | 2 (2) | 0 (0) — Change out distal locking screw
Probe misplacement (Surgical and medical procedures) | 2 (2) | 0 (0) — Probe not correctly placed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Sponsor shall have the sole right for 12 mo after completion of Study at all sites to arrange for the submission of the multi-center article or presentation
* After the 12 mo, upon Sponsor approval or after the multicenter publication occurs, Investigator may publish, present and use for instruction and research, Investigator's results arising out of its conduct of the Study at the Site. Investigator may not disclose Sponsor Confidential Information, and Sponsor protects its proprietary rights